CLINICAL TRIAL: NCT04367428
Title: Effects of Pre- and Postoperative Probiotics Administration on Postoperative Weight Loss in Patients Undergoing Sleeve Gastrectomy
Brief Title: Pre- and Postoperative Probiotics Administration in Patients Undergoing Sleeve Gastrectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Head of Bariatric Surgery Unit, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Garcilaso-Mex 2020/4
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Patients will receive the previously mentioned combination of probiotics pre- and postoperatively
  Interventions: Biological: Administration of probiotics
- No probiotics (No Intervention): Patients will not receive probiotics

INTERVENTIONS:
Biological: Administration of probiotics — Patients will receive the previously mentioned combination of probiotics before and after surgery
  Arms: Probiotics

SUMMARY:
Patients will be randomized into 2 groups:

* G1: Patients undergoing sleeve gastrectomy as bariatric procedure and receiving pre- and postoperative probiotics
* G2: Patients undergoing sleeve gastrectomy as bariatric procedure and not receiving pre- or postoperative probiotics

Weight loss will be assessed 1 year after surgery

DETAILED DESCRIPTION:
Patients will be randomized into 2 groups:

* G1: Patients undergoing sleeve gastrectomy as bariatric procedure and receiving pre- and postoperative probiotics
* G2: Patients undergoing sleeve gastrectomy as bariatric procedure and not receiving pre- or postoperative probiotics

Preoperative probiotics scheme include:

* saccharomyces boulardii ntc 5375 + enterococcus faecium UBEF-41 + lactobacillus acidophilus LA 14 during 15 days (between 6th and 4th weeks before surgery)
* Bifidobacterium lactis BL 04 + Bifidobacterium breve BB 03 + Bifidobacterium bifidum BB 06 + Bifidobacterium longum BL 05 during 15 days (between 4th and 2nd weeks before surgery)
* lactobacillus rhamnosus LR 32 + lactobacillus rhamnosus HN001 + lactobacillus acidophillus LA 14 during 15 days (between 2nd week and the day before surgery)

Postoperative probiotics scheme include:

* saccharomyces boulardii ntc 5375 + enterococcus faecium UBEF-41 + lactobacillus acidophilus LA 14 during 15 days (between 1st and 3rd weeks after surgery)
* Lactobacillus rhamnosus LR 32 + Bifidobacterium lactis BL 04 + Bifidobacterium longum BL 05 + lactobacillus salivarius LS 33 + lactobacillus acidophilus LA 14 + bifidobacterium bifidum BGN 4 during 4 months (between 4th and 20th weeks after surgery.

Both groups will receive the same nutritional recommendations.

1 year after surgery, weight los will be assessed as primary outcome. Secondary outcomes will include daibetes mellitus remission and dyslipidemia remission.

Weight loss will be assessed 1 year after surgery

ELIGIBILITY:
Inclusion Criteria:

* BMI >40
* BMI >35 associated to diabetes mellitus, hypertension, dyslipidemia or sleep apnea/hypopnea síndrome
* Patients undergoing laparoscopic sleeve gastrectomy as primary bariatric procedure

Exclusion Criteria:

* Revisional surgery
* Patients with gastroesophageal reflux disease
* Patients planned for a sleeve gastrectomy as first step of a second malabsorptive procedure
* Patients with immune deficiencies or with chronic intake of immune supressor drugs
* patients refusing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-02 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 1 year after surgery
  Weight loss will be assessed as excess body mass index (BMI) loss, calculated by the formula:
  Excess BMI loss= (preoperative BMI-postoperative BMI)/ (preoperative BMI-25)

SECONDARY OUTCOMES:
Remission of diabetes mellitus | 1 year after surgery
  Remission of diabetes mellitus will be defined as fasting glucose <100mg/dl and glycated hemoglobin <6% at blood sample
Remission of dyslipidemia | 1 year after surgery
  Remission of dyslipidemia will be defined as triglycerids <200mg/dl, total cholesterol<200mg/dl and HDL-colesterol >45mg/dl at blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Gonzalez, Study Director — Hospital Angeles del Carmen, Guadalajara, Mexico

IPD SHARING:
Plan to Share IPD: Undecided